CLINICAL TRIAL: NCT02097290
Title: CAPTure Information Via Automatic Threshold Evaluation
Brief Title: Evaluation of Automatic Threshold Algorithms
Acronym: CAPTIVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPTIVATE; IDE# G130241 (Other: FDA)
Record Dates: First submitted 2014-03-20; First posted 2014-03-27 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure
Keywords: Threshold algorithms; CRT-D
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRT-D (Experimental): For all subjects with the AUTOGEN CRT-D, the autothreshold algorithms will be evaluated
  Interventions: Device: CRT-D

INTERVENTIONS:
Device: CRT-D — For all subjects with the AUTOGEN CRT-D, the autothreshold algorithms will be evaluated

SUMMARY:
This study will evaluate the PaceSafe Right Ventricular Autothreshold (RVAT) and Left Ventricular Autothreshold (LVAT) features for AUTOGEN Cardiac Resynchronization Therapy Defibrillator (CRT-D) devices.

DETAILED DESCRIPTION:
The objective of the CAPTIVATE Clinical Study is to gather data to establish the safety and effectiveness of the PaceSafe Right Ventricular Autothreshold (RVAT) and Left Ventricular Autothreshold (LVAT) features to support the regulatory approval of the AUTOGEN CRT-D family of devices.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects prescribed a CRT-D and indicated per guidelines, who will receive an AUTOGEN CRT-D model G160, G161, G172, G173
2. Subjects who have an implanted functional endocardial right ventricular defibrillation lead or who will receive a endocardial right ventricular defibrillation lead
3. Subjects who have an implanted functional bipolar or unipolar left ventricular lead or who will receive a bipolar or unipolar left ventricular lead
4. Subjects who are willing and capable of providing informed consent to undergo a device implant procedure, and to participate in all testing and follow-ups defined in this protocol
5. Subjects whose age is 18 or above, or of legal age to give informed consent specific to national law

Exclusion Criteria:

1. Subjects who have an implanted multipolar (>2poles) left ventricular lead or who will receive a multipolar (>2poles) left ventricular lead
2. Subjects with an unknown model/manufacturer, or implant date for the RA, RV or LV lead
3. Subjects for whom a RV defibrillation lead manufactured by St. Jude Medical or Biotronik is implanted, is planned to be implanted, or has been abandoned
4. Implanted with an active Medtronic Sprint Fidelis® lead models: 6930, 6931, 6948 or 6949
5. Subjects with an implanted or abandoned St. Jude Medical QuickSite® or QuickFlex® lead models: 1056T, 1058T, 1156T, 1158T
6. Subjects with a RV or LV lead revision or extraction within 30 days of enrollment
7. Subjects with an implanted lead that is planned to be extracted during the study implant procedure
8. Subjects with an active implanted RA or RV lead that is greater than 10 years old, unless the lead will be abandoned
9. Subjects with an active implanted LV lead that is greater than 8 years old, unless the lead will be abandoned
10. Subjects preexisting unipolar pacemaker that will not be explanted/abandoned
11. Subjects with a life expectancy less than 6 months
12. Subjects with a prosthetic mechanical tricuspid heart valve
13. Women of childbearing age who are pregnant or plan to become pregnant. NOTE: women of childbearing potential with an uncertain pregnancy status must have a negative pregnancy test within 7 days prior to enrollment. Pregnancy tests are required as part of standard routing clinical practice at all centers whenever female patients are exposed to x-ray radiation. Since this protocol does not require any exposure of the female patients to x-ray and x-ray exposure is part of the clinical procedure, it is the responsibility of the investigators to ensure that pregnant females will not be exposed to x-ray at any time
14. Subject enrolled in a concurrent study, except national/governmental registries that do not require a signed informed consent form, without the written approval from Boston Scientific
15. Subjects who are not geographically stable, to the extent that it would prevent attending the study follow-ups at the investigational center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ellenbogen, MD, Principal Investigator — Virginia Commonwealth University Medical Center
Locations (36):
- United States (36):
  - Glendale Adventist Medical Center, Glendale, California
  - Danbury Hospital, Danbury, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Delray Medical Center, Atlantis, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - First Coast Cardiovascular, Jacksonville, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - University Community Hospital, Trinity, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Carle Foundation Hospital, Urbana, Illinois
  - IU Health LaPorte, La Porte, Indiana
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - University of Iowa Hospitals and Clinics, Davenport, Iowa
  - Via-Christi Regional Medical Center, Wichita, Kansas
  - Norton Cardiovascular Associates, Louisville, Kentucky
  - University of Maryland Medical System, Baltimore, Maryland
  - Steward St. Elizabeth's Medical Center of Boston, Inc., Boston, Massachusetts
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Sparrow Health System, Lansing, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Cox Health, Springfield, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Rochester General Hospital, Rochester, New York
  - Wake Medical Center, Raleigh, North Carolina
  - Summa Health System, Akron, Ohio
  - Lindner Center for Research and Education, Cincinnati, Ohio
  - St. Elizabeth Health Center, Poland, Ohio
  - Good Samaritan Hospital, Lebanon, Pennsylvania
  - University Medical Center-Greenville Memorial Hospital, Greenville, South Carolina
  - Seton Medical Center, Austin, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - Virginia Commonwealth University Health, Richmond, Virginia
  - PeaceHealth Southwest Medical, Vancouver, Washington
  - St. Mary's Medical Center, Huntington, West Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRT-D
Started | 210
Completed | 193 (Active subjects at the end of 3 month follow up visit for primary end point data collection)
Not Completed | 17
Not completed — Death | 6
Not completed — Total Withdrawals | 3
Not completed — Attempt | 8

BASELINE CHARACTERISTICS:
Arm/Group | CRT-D
Number analyzed (Participants) | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 8
  Multiple Races | 3
  Asian | 1
  Black | 25
  Other | 1
  White | 170
  Undisclosed | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 210

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint is to Evaluate the System-related Complication-free Rate
Description: Safety of the AUTOGEN was evaluated by the system-related complication-free rate (CFR) at 3-months post-implant. The system consists of the implanted AUTOGEN CRT-D pulse generator, RA lead (if implanted), RV lead, and LV lead.
Time Frame: 3 months
Population: Implant + Attempt Subjects
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CRT-D
Number analyzed (Participants) | 210
Percentage of participants | 84.2 [79.5 to NA] — Only lower confidence interval limit was considered for end point result

2. Primary Outcome: The Accuracy of the RVAT Commanded Test Will be Evaluated by Comparing the RVAT Determined Threshold to a Core Lab (Independent Physician) Determined Threshold.
Description: Accuracy of the algorithm will be measured for all patients, by comparing algorithm determined threshold to a core lab determined threshold at both the 1-month and 3-month follow-up visits. The RVAT determined threshold for all patients at 1-month and 3-month follow-up visits are pooled for final analysis. An accurate commanded threshold is defined by: |commanded threshold - core lab determined threshold| ≤ 0.2 V; if the commanded threshold is ≤ 3.5V or |commanded threshold - core lab determined threshold| ≤ 0.5 V; if the commanded threshold is > 3.5V. Subjects were allowed to contribute multiple paired datasets for this endpoint analysis, one set each from the 1-month and 3-month visits. Paired datasets from the 1-month and 3-month visits were pooled for the purpose of this endpoint analysis.
Time Frame: 1-month and 3-month follow-up visits
Population: A total of 288 paired datasets (from 171 unique subjects in whom RVAT threshold was available), each dataset consisting of a commanded RVAT threshold and a core lab determined threshold, were collected at the 1-month and 3- month visits and pooled for final analysis.
Measure: Number (95% Confidence Interval); unit: percentage of commanded RVAT thresholds
Units Other Than Participants: Commanded RVAT thresholds paired dataset
Arm/Group | CRT-D
Number analyzed (Participants) | 171
Number analyzed (Commanded RVAT thresholds paired dataset) | 288
percentage of commanded RVAT thresholds | 97.9 [95.9 to NA] — Only lower confidence interval limit was considered for end point result

3. Primary Outcome: The Accuracy of the LVAT Commanded Test Will be Evaluated by Comparing the LVAT Determined Threshold to a Core Lab (Independent Physician) Determined Threshold.
Description: Accuracy of the algorithm will be measured for all patients, by comparing algorithm determined threshold to a core lab determined threshold at both the 1-month and 3-month follow-up visits. The LVAT determined threshold for all patients at 1-month and 3-month follow-up visits are pooled for final analysis. An accurate commanded threshold is defined by: commanded threshold - core lab determined threshold| ≤ 0.2 V; if the commanded threshold is ≤ 3.5V or |commanded threshold - core lab determined threshold| ≤ 0.5 V; if the commanded threshold is > 3.5V. Paired datasets from the 1-month and 3-month visits were pooled for the purpose of this endpoint analysis. Subjects were allowed to contribute multiple paired datasets for this endpoint analysis, one set each from the 1-month and 3-month visits. Paired datasets from the 1-month and 3-month visits were pooled for the purpose of this endpoint analysis.
Time Frame: 1-month and 3-month follow up visits
Population: A total of 324 paired datasets (from 182 unique subjects in whom LVAT threshold was available), each dataset consisting of a commanded LVAT threshold and a core lab determined threshold, were collected at the 1-month and 3- month visits and pooled for final analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of commanded LVAT thresholds
Units Other Than Participants: Commanded LVAT thresholds-paired dataset
Arm/Group | CRT-D
Number analyzed (Participants) | 182
Number analyzed (Commanded LVAT thresholds-paired dataset) | 324
Percentage of commanded LVAT thresholds | 97.8 [96.0 to NA] — Only lower confidence interval limit was considered for end point result

4. Primary Outcome: The Accuracy of the RVAT Ambulatory Test Will be Evaluated by Comparing the RVAT Determined Threshold to a Core Lab (Independent Physician) Determined Threshold
Description: Accuracy of the algorithm will be measured for all patients, by comparing algorithm determined threshold to a core lab determined threshold at both the 1-month and 3-month follow-up visits.The RVAT determined threshold for all patients at 1-month and 3-month follow-up visits are pooled for final analysis. An accurate Ambulatory threshold is defined by:|Ambulatory threshold - ECG threshold| ≤ 0.6 V; if the ECG threshold is ≤ 3.5V or |Ambulatory threshold - ECG threshold| ≤ 1.0 V; if the ECG threshold is > 3.5V. Subjects were allowed to contribute multiple paired datasets for this endpoint analysis, one set each from the 1-month and 3-month visits. Paired datasets form the 1-month and 3-month visits were pooled for purposes of endpoint analysis.
Time Frame: 1-month and 3-month follow up visits
Population: A total of 314 paired datasets (from 183 unique subjects in whom RVAT threshold was available), each dataset consisting of an ambulatory RVAT threshold and a core lab determined threshold, were collected at the 1-month and 3- month visits and pooled for final analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of RVAT ambulatory thresholds
Units Other Than Participants: RVAT ambulatory threshold paired dataset
Arm/Group | CRT-D
Number analyzed (Participants) | 183
Number analyzed (RVAT ambulatory threshold paired dataset) | 314
Percentage of RVAT ambulatory thresholds | 99.0 [97.5 to NA] — Only lower confidence interval limit was considered for end point result

5. Primary Outcome: The Accuracy of the LVAT Ambulatory Test Will be Evaluated by Comparing the LVAT Determined Threshold to a Core Lab (Independent Physician) Determined Threshold
Description: Accuracy of the algorithm will be measured for all patients, by comparing algorithm determined threshold to a core lab determined threshold at both the 1-month and 3-month follow-up visits. The LVAT determined threshold for all patients at 1-month and 3-month follow-up visits are pooled for final analysis. An accurate Ambulatory threshold is defined by: |Ambulatory threshold - ECG threshold| ≤ 1.0 V. Paired datasets from the 1-month and 3-month visits were pooled for the purpose of this endpoint analysis. Subjects were allowed to contribute multiple paired datasets for this endpoint analysis, one set each from the 1-month and 3-month visits. Paired datasets form the 1-month and 3-month visits were pooled for purposes of endpoint analysis.
Time Frame: 1-month and 3-month follow up visits
Population: A total of 300 paired datasets (from 175 unique subjects in whom LVAT threshold was available), each dataset consisting of a ambulatory LVAT threshold and a core lab determined threshold, were collected at the 1-month and 3- month visits and pooled for final analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of accurate threshold
Units Other Than Participants: LVAT ambulatory threshold paired dataset
Arm/Group | CRT-D
Number analyzed (Participants) | 175
Number analyzed (LVAT ambulatory threshold paired dataset) | 300
Percentage of accurate threshold | 97.7 [95.7 to NA] — Only lower confidence interval limit was considered for end point result

6. Secondary Outcome: RVAT Secondary Efficacy Endpoint: The Percent of RVAT Commanded Tests That Result in an Appropriate Outcome
Description: This endpoint will evaluate the percent of RVAT commanded tests that result in an appropriate outcome. There are three possible outcomes to a commanded test:
  1. A device-determined threshold
  2. A threshold test code (indicating that a threshold could not be determined) representing an error condition that is beyond the control of the RVAT feature and could occur in the manual threshold tests
  3. A threshold test code (indicating that a threshold could not be determined) that was due to a limitation of the RVAT feature and might not occur in manual threshold tests An appropriate RVAT outcome consists of the first two outcomes listed above: a device-determined threshold and a threshold test code representing an error condition that is beyond the control of the RVAT feature and could occur in the manual threshold tests. An inappropriate RVAT outcome consists of the last of the three outcomes listed above.
Time Frame: 3-month follow up visit
Population: A total of 157 unique subjects in whom a paired RVAT dataset was collected at the 3-month follow up visit. A paired dataset consisted of an RVAT threshold test outcome and core lab determined threshold test outcome.
Measure: Number (95% Confidence Interval); unit: percentage of appropriate outcome
Arm/Group | CRT-D
Number analyzed (Participants) | 157
percentage of appropriate outcome | 85.4 [79.9 to NA] — Only lower confidence interval limit was considered for end point result

7. Secondary Outcome: LVAT Secondary Efficacy Endpoint: The Percent of LVAT Commanded Tests That Result in an Appropriate Outcome
Description: This endpoint will evaluate the percent of LVAT commanded tests that result in an appropriate outcome. There are three possible outcomes to a commanded test:
  1. A device-determined threshold
  2. A threshold test code (indicating that a threshold could not be determined) representing an error condition that is beyond the control of the LVAT feature and could occur in the manual threshold tests
  3. A threshold test code (indicating that a threshold could not be determined) that was due to a limitation of the LVAT feature and might not occur in manual threshold tests An appropriate LVAT outcome consists of the first two outcomes listed above: a device-determined threshold and a threshold test code representing an error condition that is beyond the control of the LVAT feature and could occur in the manual threshold tests. An inappropriate LVAT outcome consists of the last of the three outcomes listed above.
Time Frame: 3-month follow up visit
Population: A total of 182 unique subjects in whom a paired LVAT dataset was collected at the 3-month follow up visit. A paired dataset consisted of an LVAT threshold test outcome and core lab determined threshold test outcome.
Measure: Number (95% Confidence Interval); unit: percentage of appropriate outcome
Arm/Group | CRT-D
Number analyzed (Participants) | 182
percentage of appropriate outcome | 95.1 [91.5 to NA] — Only lower confidence interval limit was considered for end point result

ADVERSE EVENTS:
Time Frame: Adverse events reported were collected from ICF signature until the last study follow-up.
Groups:
- CRT-D: CRT-D: For all subjects with the AUTOGEN CRT-D, the autothreshold algorithms will be evaluated.
  Subjects in whom AUTOGEN CRT-D was successfully implanted or an attempt to implant made were considered to be at risk for adverse events. There were a total of 210 implants and attempts.
Arm/Group | CRT-D
All-Cause Mortality (participants affected / at risk) | 17/210
Serious Adverse Events (participants affected / at risk) | 101/210
Other Adverse Events (participants affected / at risk) | 81/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-D (N=210)
Abnormal Laboratory Values (Blood and lymphatic system disorders) | 2 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
Adverse Reaction - Hypotension (Cardiac disorders) | 2 (2)
Adverse Reaction - Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Arterial/Venous Trombolytic Event (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Af) (Cardiac disorders) | 7 (8)
Atrial Flutter (Cardiac disorders) | 5 (5)
Atrial Tachyarrhythmias (Cardiac disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Cardiac Arrest (Cardiac disorders) | 8 (8)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cerebrovascular Accident (Cva) (Vascular disorders) | 1 (1)
Chest Pain - Ischemic (Cardiac disorders) | 3 (3)
Chest Pain - Other (Cardiac disorders) | 3 (3)
Copd Exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Coronary Artery Disease (Cardiac disorders) | 1 (2)
Coronary Venous Perforation Without Tamponade (Cardiac disorders) | 1 (1)
Dislodgment - Elevated Threshold - Rv (Cardiac disorders) | 1 (1)
Dislodgment - Extracardiac Stimulation - Lv (Cardiac disorders) | 1 (1)
Dislodgment - Multiple Signs - Rv (Cardiac disorders) | 1 (2)
Dislodgment - No Reported Signs - Lv (Cardiac disorders) | 3 (3)
Dislodgment - No Reported Signs - Ra (Cardiac disorders) | 1 (1)
Dislodgment - Unable To Capture - Lv (Cardiac disorders) | 3 (3)
Dislodgment - Unable To Capture - Ra (Cardiac disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Dyspnea - Heart Failure (Cardiac disorders) | 9 (13)
Elevated Threshold - Lv (Cardiac disorders) | 1 (1)
Endocrine (Endocrine disorders) | 4 (5)
Extracardiac Stimulation - Lv (Cardiac disorders) | 5 (5)
Gastrointestinal (Gastrointestinal disorders) | 14 (17)
Gastrointestinal - Heart Failure (Cardiac disorders) | 1 (1)
Genitourinary (Renal and urinary disorders) | 7 (7)
Cataract (Eye disorders) | 2 (2)
Heart Failure Symptoms - Unspecified (Cardiac disorders) | 6 (6)
Hematological (Blood and lymphatic system disorders) | 4 (5)
Hematoma - Pocket (<=30 Days Post-Implant) (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Cardiac disorders) | 2 (2)
Hypotension - Heart Failure (Cardiac disorders) | 1 (1)
Impedance < 300 Ohms - Ra (Cardiac disorders) | 1 (1)
Inadvertent Vt/Vf (Cardiac disorders) | 1 (1)
Inappropriate Tachy Therapy - Svt (Cardiac disorders) | 2 (2)
Infection (> 3 Days Post-Implant) (Infections and infestations) | 1 (1)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 1 (1)
Migration (Ear and labyrinth disorders) | 1 (1)
Mitral Regurgitation (Cardiac disorders) | 1 (1)
Multi-System Failure (Immune system disorders) | 1 (1)
Multi-System Failure - Heart Failure (Cardiac disorders) | 5 (5)
Multiple Heart Failure Symptoms (Cardiac disorders) | 25 (34)
Multiple Symptoms (Immune system disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (6)
Myocardial Infarction (Cardiac disorders) | 4 (4)
Myocardial Perforation Post-Implant - Rv (Cardiac disorders) | 1 (1)
Myocardial Perforation With Tamponade (Cardiac disorders) | 1 (1)
Neurological (Nervous system disorders) | 4 (5)
Other-Lead-Procedure (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 2 (2)
Peripheral Edema - Heart Failure (Cardiac disorders) | 1 (1)
Peripheral Vascular Disease (Vascular disorders) | 3 (3)
Physical Trauma (Musculoskeletal and connective tissue disorders) | 3 (3)
Pleural Effusion (Cardiac disorders) | 1 (2)
Pneumothorax - Procedure (Cardiac disorders) | 4 (4)
Post-Surgical Wound Discomfort (Skin and subcutaneous tissue disorders) | 2 (2)
Premature Ventricular Contractions (Pvc) (Cardiac disorders) | 1 (1)
Psychological (Psychiatric disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 14 (23)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Edema - Heart Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal (Renal and urinary disorders) | 7 (8)
Renal Failure Due To Contrast Media - Procedure (Renal and urinary disorders) | 1 (1)
Renal Insufficiency - Heart Failure (Renal and urinary disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 3 (3)
Systemic Infection (Infections and infestations) | 4 (5)
Unable To Capture - Lv (Cardiac disorders) | 1 (1)
Unable To Convert - Defibrillation (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Vf) (Cardiac disorders) | 2 (2)
Ventricular Flutter (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Vt) (Cardiac disorders) | 3 (4)
Failure To Implant Epicardial Lv Lead (Cardiac disorders) | 1 (1)
Inability To Place The Lv Lead (Cardiac disorders) | 1 (1)
Left Chest Wall Emphysema (Cardiac disorders) | 1 (1)
Left Leg Ischemia (Vascular disorders) | 1 (1)
ICD shocks (Cardiac disorders) | 2 (2)
Severe Rt. Leg Stump Infection (Infections and infestations) | 1 (1)
Unable To Insert Lv Lead With Initial Procedure (Cardiac disorders) | 1 (1)
Vestibulitis (Ear and labyrinth disorders) | 1 (1)
Angioedema (General disorders) | 1 (1)
Patient Death - unknown cause (General disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT-D (N=210)
Abnormal Laboratory Values (General disorders) | 7 (10)
Allergic Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Delirium (General disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 11 (12)
Atrial Flutter (Cardiac disorders) | 3 (3)
Atrial Tachyarrhythmias (Cardiac disorders) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Unable to perform Threshold test-RV (Cardiac disorders) | 1 (1)
Chest Pain-Ischemic (Cardiac disorders) | 1 (1)
Chest Pain-Other (Cardiac disorders) | 5 (5)
COPD (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Coronary Venous Dissection (Cardiac disorders) | 2 (2)
Dislodgment-extracardiac stimulation-RA (Cardiac disorders) | 1 (1)
Dislodgment-LV (Cardiac disorders) | 1 (1)
Dislodgment-unable to capture-LV (Cardiac disorders) | 1 (1)
Dislodgment-unable to capture-RV (Cardiac disorders) | 1 (1)
Dizziness (General disorders) | 4 (4)
Dyspnea-heart failure (Cardiac disorders) | 3 (3)
Endocrine (Endocrine disorders) | 5 (5)
Extracardiac stimulation-LV (Cardiac disorders) | 28 (30)
Fatigue (General disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 8 (10)
Genitorurinary (Renal and urinary disorders) | 10 (11)
Visual disturbances (Eye disorders) | 2 (3)
Hematological (Blood and lymphatic system disorders) | 6 (6)
Hematoma (less than 30 days post implant) (Skin and subcutaneous tissue disorders) | 7 (7)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Immune disorder (Immune system disorders) | 1 (1)
Insulation breach-RV (Cardiac disorders) | 1 (1)
Integumentary (Skin and subcutaneous tissue disorders) | 8 (8)
Mitral regurgitation (Cardiac disorders) | 1 (1)
Multiple Heart Failure Symptoms (Cardiac disorders) | 5 (7)
Muskuloskeletal (Musculoskeletal and connective tissue disorders) | 14 (16)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Neurological (Nervous system disorders) | 3 (4)
Nonsustained Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Other PG-system-procedure (Cardiac disorders) | 1 (1)
Cardiovascular event (Cardiac disorders) | 1 (1)
Oversensing-RV (Cardiac disorders) | 1 (1)
Pacemaker Mediated Tachycardia (Cardiac disorders) | 8 (8)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral edema-heart failure (Cardiac disorders) | 2 (2)
Peripheral vascular disease (Vascular disorders) | 1 (1)
PG system-event (Cardiac disorders) | 1 (1)
Physical Trauma (Musculoskeletal and connective tissue disorders) | 11 (12)
Post surgical infection (Infections and infestations) | 1 (1)
Post-surgical Pocket Hemorhage (Skin and subcutaneous tissue disorders) | 1 (1)
Post-surgical wound discomfort (Skin and subcutaneous tissue disorders) | 9 (9)
Premature ventricular contractions (Cardiac disorders) | 1 (1)
Psychological (Psychiatric disorders) | 2 (3)
Psychological effect due to device therapy (Psychiatric disorders) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Renal (Renal and urinary disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Thromboembolic events (Cardiac disorders) | 1 (1)
Transient Ischemic Attack (Cardiac disorders) | 1 (1)
Unable to capture-LV lead (Cardiac disorders) | 2 (2)
Undersensing-RA (Cardiac disorders) | 1 (1)
Venous Occlusion (Vascular disorders) | 1 (1)
Ventricular Tacchyarrhythmias (Cardiac disorders) | 1 (1)
Weight Gain (General disorders) | 1 (1)
Adverse Drug Reaction (General disorders) | 1 (1)
Cocaine Abuse (General disorders) | 1 (1)
Ear reaction (Ear and labyrinth disorders) | 1 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Swollen neck (Skin and subcutaneous tissue disorders) | 1 (1)
ICD shocks (Cardiac disorders) | 1 (1)
Low LVEF (Cardiac disorders) | 1 (1)
High LV lead impedance (Cardiac disorders) | 1 (1)
High RV lead impedance (Cardiac disorders) | 1 (1)
Low pacing output (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The RVAT and LVAT endpoints are compared against a performance goal rather than to a randomized control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days